CLINICAL TRIAL: NCT03810391
Title: Using Preoperative Anxiety Score to Determine the Total Dose of Butorphanol for Sedation in Patients Undergoing Lower Limb Orthopedic Procedures: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Using Preoperative Anxiety Score to Determine the Total Dose of Butorphanol for Sedation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Effect of butorphanol
Record Dates: First submitted 2019-01-13; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Preoperative Anxiety Score; Total Dose of Butorphanol
Keywords: Butorphanol; preoperative anxiety; sedation; recommend dose
MeSH Terms: interventions — Butorphanol

STUDY DESIGN:
Intervention Model Description: the Amsterdam preoperative anxiety and information scale was used to evaluated the degree of preoperative anxiety one day before the surgery. Patients in preoperative anxiety group were randomly allocated to two groups: butorphanol group (Group A) and physiological saline group (Group B); Patients in non-preoperative anxiety group were also randomly allocated to two groups: butorphanol group (Group C) and physiological saline group (Group D) In Group A and Group C, patients received an intravenous loading dose of 15ug/kg butorphanol 5 mins before starting the surgery, then followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion when the Ramsay sedation score (RSS) reached 4 , Group B and Group D received an infusion of the same volume of physiological saline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- preoperative anxiety and butorphanol (Experimental): preoperative anxiety scores of patients in Group A were >11 and received an intravenous loading dose of 15ug/kg butorphanol 5 min before starting the surgery, then followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion until the Ramsay sedation score reached 4 points
  Interventions: Drug: Butorphanol
- preoperative anxiety and saline (Placebo Comparator): preoperative anxiety scores of patients in Group B were >11 and received an infusion of the same volume of physiological saline
  Interventions: Other: physiological saline
- non-preoperative anxiety and butorphanol (Experimental): preoperative anxiety scores of patients in Group C were ≤ 11 and received an intravenous loading dose of 15ug/kg butorphanol 5 min before starting the surgery, then followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion until the Ramsay sedation score reached 4 points
  Interventions: Drug: Butorphanol
- non-preoperative anxiety and saline (Placebo Comparator): preoperative anxiety scores of patients in Group D were ≤11 and received an infusion of the same volume of physiological saline
  Interventions: Other: physiological saline

INTERVENTIONS:
Drug: Butorphanol — intravenous loading dose of 15ug/kg butorphanol,and followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion until the Ramsay sedation score reached 4 points
  Other Names: butorphanol tartrate injection
  Arms: non-preoperative anxiety and butorphanol; preoperative anxiety and butorphanol
Other: physiological saline — intravenous infusion of the same volume of physiological saline
  Arms: non-preoperative anxiety and saline; preoperative anxiety and saline

SUMMARY:
Orthopedic surgeries are considered to be discomfortable and the sense of fear and anxiety of patients who already have preoperative anxiety may be aggravated by intraoperative stimulation, which may contribute to postoperative complications. Previous studies have found that high anxiety predicts increased sedative requirements. Therefore, the investigators explored the relationship between anxiety and intraoperative butorphanol requirements and the investigators evaluated the specific sedative requirement which can keep satisfactory sedative state for patients by preoperative anxiety score

DETAILED DESCRIPTION:
A total of one hundred and eighteen patients who were to undergoing lower limb orthopedic procedures with spinal anesthesia were selected，the Amsterdam preoperative anxiety and information scale was used to evaluated the degree of preoperative anxiety one day before the surgery. Patients in preoperative anxiety group were randomly allocated to two groups: butorphanol group (Group A) and physiological saline group (Group B); Patients in non-preoperative anxiety group were also randomly allocated to two groups: butorphanol group (Group C) and physiological saline group (Group D). In Group A and Group C, patients received an intravenous loading dose of 15ug/kg butorphanol 5 min before starting the surgery, then followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion until the Ramsay sedation score reached 4 points, Group B and Group D received an infusion of the same volume of physiological saline. The sedation scores were recorded 10 min after getting into the operation room and 5, 10, 15, 30min after infusion of butorphanol or physiological saline. The duration when Ramsay sedation score reached 4 points in Group A and C, adverse events and post-operative visual analgesia scale scores were also recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA)Ⅰ-Ⅱ
* 18-75 years
* Scheduled for elective low limb orthopaedic procedures under spinal anesthesia

Exclusion Criteria:

* central system disease
* cardiovascular disease
* autonomic nervous system disease
* long term use of analgesic, sedative, and anti-anxiety drugs
* psychosis
* a patient with a language communication disorder not willing to cooperate with the experimenter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
preoperative anxiety score (Amsterdam preoperative anxiety and information scale, APAIS) | one day before the surgery
  evaluate the preoperative anxiety score one day before the surgery, the scale ranges from 0-33. And we define a score of 11 as a cut-off point, the higher the score the more serious the preoperative anxiety is
Ramsay sedation score (Ramsay sedation scale, RSS) | during the surgery
  evaluate the Ramsay sedation score 10 min after getting into the operation room and 5, 10, 15, 30min after infusion. The Ramsay sedation scale ranges from 1-6. 1, anxious and agitated or restless or both; 2, cooperative, orientated, and tranquil; 3, responds to commands only; 4, brisk response to a light glabellar tap or auditory stimulus; 5, sluggish response to a light glabellar tap or auditory stimulus; and 6, no response to a light glabellar tap or auditory stimulus. A sedative state with RSS 4 was considered as an adequate level of sedation
the time when Ramsay sedation score reached 4 points | Ramsay sedation score reach 4 points during the surgery
  record the time when Ramsay sedation score reached 4 points. The Ramsay sedation scale ranges from 1-6. 1, anxious and agitated or restless or both; 2, cooperative, orientated, and tranquil; 3, responds to commands only; 4, brisk response to a light glabellar tap or auditory stimulus; 5, sluggish response to a light glabellar tap or auditory stimulus; and 6, no response to a light glabellar tap or auditory stimulus. A sedative state with RSS 4 was considered as an adequate level of sedation

SECONDARY OUTCOMES:
vital signs | during the surgery
  Record Mean Arterial Pressure(MAP)10 min after getting into the operation room and 5, 10, 15, 30min after infusion
The incidence of nausea/ vomiting, dizzy, bradycardia and hypotension | in the first day after the surgery
  Investigate the incidence of nausea/ vomiting, dizzy, bradycardia and hypotension in the first day after the surgery
post-operative visual analgesia scale scores (VAS) | within 24 hours after the surgery
  investigate the VAS every hour till 6 hours and then every 2 hours till 24 hours. The VAS ranges from 1-10. 0 means painless; 1-3 means mild pain; 4-6 means moderate pain and 7-10 means severe pain
Vital signs | during the surgery
  Record Spo2 10 min after getting into the operation room and 5, 10, 15, 30min after infusion
Vital signs | during the surgery
  Record Heart Rate(HR) 10 min after getting into the operation room and 5, 10, 15, 30min after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, professor, Study Director — Shengjing Hospital
Locations (1):
- shengjing hospital of China medical university, Shenyang, Liaoning, China